CLINICAL TRIAL: NCT03145272
Title: Pharmacokinetics and Pharmacogenomics of Oral Oxycodone in Thai Pediatric Surgical Patients : a Pilot Study
Brief Title: Population Pharmacokinetics and Pharmacogenomics of Oral Oxycodone in Thai Pediatric Surgical Patients
Acronym: PedPK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI407/2016
Record Dates: First submitted 2017-04-24; First posted 2017-05-09 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Pharmacokinetics; Pharmacogenomics; Oxycodone
Keywords: Pharmacogenomics; Pharmacokinetics; Oxycodone
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Age group (Experimental): An orogastric tube will be placed in the stomach (placement verified by routine accepted clinical guidelines) under anesthesia as is part of standard routine clinical care to remove gastric contents. The same orogastric tube will be used for intragastric liquid oxycodone administration in a dose of 0.1 mg/kg before the surgical incision. This weight-adjusted dose of 0.1 mg/kg is administered as per standard clinical dosing guidelines.
  This arm can be divided into 2 subgroups; (1)12 months - 1.9 years age group. (2) 2 - 5.9 years age group.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — A single weight-adjusted oxycodone dose of 0.1 mg/kg is administered as per standard clinical dosing guidelines

SUMMARY:
This study is designed as an experimental trial which collect prospective data at Mahidol university. It aims to characterize the responses of Thai pediatric population,age 1 - 6 years, to oxycodone oral syrup and its metabolites (oxymorphone, noroxymorphone and noroxycodone) with specific respect to the pharmacogenomics (How drug affects patients).

A total of 20 generally healthy, opioid-naive children, aged 1-6 years, scheduled as in-patient surgery for non-emergency surgery, non-gastrointestinal tract surgery are involved.

The patients are divide into 2 groups (1) 10 patients in 12 months - 1.9 years, and (2) 10 patients in the 2 - 5.9 years age group.

Every patient will receive inhalational or intravenous induction of anesthesia as decided by the anesthesia team on the day of surgery, as is routine clinical care. An intravenous cannula (IV) will be inserted in every patient as part of their routine clinical care. No additional intravenous line will be required for this study.

As part of the study protocol, a blood sample (5 mL) will be taken from the IV and sent for genetic analysis. (However, in order to limit the amount of blood drawn from small babies, 3 ml will be drawn, not 5 ml, if the patient is less than 6 months or less than 10kg.) The genetic testing is specifically to analyze the following genotypes only: CYP2D6 and CYP3A4, which represent the differences in cytochrome P450 metabolism of oxycodone.

An orogastric tube will be placed in the stomach under anesthesia as is part of standard routine clinical care to remove gastric contents. The same orogastric tube will be used for intragastric liquid oxycodone administration in a dose of 0.1 mg/kg before the surgical incision. This weight-adjusted dose of 0.1 mg/kg is administered as per standard clinical dosing guidelines. 10 blood samples (51mL/sample) will be taken from the IV and sent for drug-level analysis. A total of 11 blood samples will be drawn for the study. The first sample will be sent for genetic testing. The other 10 samples will be drawn at the following time points: 30 minutes, 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose in every patient and the other 2 samples anytime between 6 and 24 hours post-dose .

Oxycodone, oxymorphone, noroxymorphone and noroxycodone levels, at 10 time points, will be used to determine the individual responses to oxycodone. CYP2D6 genotype will be determined to identify the ultra-rapid metabolizers.

DETAILED DESCRIPTION:
Oxycodone is the most commonly used analgesic for the management of moderate and severe postoperative pain. The efficacy of Oxycodone as a potent opioid has been confirmed in children.

The principal metabolic pathway of oxycodone in humans is N-demethylation via enzyme CYP3A4 to generate inactive noroxycodone. A smaller amount (approximately 11%) is O-demethylated by cytochrome P450 enzyme CYP2D6 to become oxymorphone, the active and potent metabolite which exhibits about 40 times the affinity and 8 times the potency on μ-opioid receptors compared to the mother substance. Approximate frequencies of cytochrome P450 enzyme CYP2D6 phenotypes for the Caucasian population are: poor metabolizers 5 - 10%, extensive/intermediate metabolizers 65-90%, and ultra-rapid metabolizers 5 - 10%. Kirchheiner and colleagues noticed more codeine-related sedative side-effects in ultra-rapid metabolizers. In studies investigating extensive and poor metabolizers, codeine side-effects do not seem to be related to CYP2D6 genotype. However, clinical investigations of CYP2D6 genotype in the postoperative pain setting have shown conflicting results, and well-designed prospective studies are lacking. Taken together, these results demonstrate the need for careful pharmacokinetic studies in children who received a pharmacologic agent, such as oxycodone, which is metabolized by the enzyme CYP2D6.

The population PK of oxycodone and its metabolites has not been fully established for oral oxycodone in pediatric patients. In addition, there is a group of ultra-rapid metabolizers (approximately 4.5% of the population, but as high as 20% in some particular ethnic groups; East African and Saudi Arabian populations) which may be at risk for serious side effects in the commonly prescribed dose (which is extrapolated from adult recommendations). It is important to further investigate oral oxycodone to optimize dosing recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient who scheduled for non-emergency surgery
* Aged between 1 - 6 years
* Healthy volunteer
* Body weight more than 4.5 kilograms
* Opioid naive
* Schedule for pediatric non- GI tract surgery

Exclusion Criteria:

* Currently taking CYP 3A4 or CYP 2D6 inhibitors/inducers
* Known history of allergy to oxycodone
* Known GI, hepatic, or renal dysfunction
* Known sleep apnea or impaired respiratory reserve

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics metric (serum level of oxycodone and its metabolites at different time points) | Up to 24 hours
  Oxycodone, oxymorphone, noroxymorphone and noroxycodone serum levels [ Time Frame: The 10 samples will be drawn at the following time points: 8 blood samples will be taken at 30 minutes, 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose in every patient along other 2 samples at approximately either 8 and 12 or 10 and 24 hours post-dose. ] Oxycodone, oxymorphone, noroxymorphone and noroxycodone levels in blood (ng/ml), at 10 time points, will be used to determine the effects of single-dose oral oxycodone administration in children.

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Srisawasdi, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No